CLINICAL TRIAL: NCT02242799
Title: Evaluation of Dolutegravir Interactions With Artemether-Lumefantrine and Amodiaquine-Artesunate
Brief Title: Dolutegravir Interactions With Artemisinin-based Combination Therapies
Acronym: DolACT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Liverpool (Other)
Collaborators: ViiV Healthcare (Industry); Makerere University (Other)
Responsible Party: Principal Investigator, Catriona Waitt, Site sub-investigator, University of Liverpool
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PK13
Record Dates: First submitted 2014-09-13; First posted 2014-09-17 (Estimated); Last update posted 2016-10-05 (Estimated); Status verified 2016-10

CONDITIONS: Malaria; HIV
Keywords: Malaria; HIV; Dolutegravir; Artemisinin; Pharmacokinetics; Interactions
MeSH Terms: conditions — Malaria | interventions — dolutegravir; Artemether, Lumefantrine Drug Combination; amodiaquine, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Study A Sequence 1 (Experimental): Artemether-lumefantrine combination alone for 3 days with PK sampling at steady state, then 21 day washout period followed by Dolutegravir 50mg od dosing to steady state (7 days) with PK sampling then a further 3 days where Artemether-lumefantrine combination and Dolutegravir 50mg od are given together, with PK sampling at steady state.
  Interventions: Drug: Dolutegravir 50mg od; Drug: Artemether-lumefantrine combination
- Study A Sequence 2 (Experimental): Dolutegravir 50mg od given for 7 days with PK sampling at steady state, followed immediately by a further 3 days where Artemether-lumefantrine combination and Dolutegravir 50mg od are given together, again with PK sampling at steady state. Following a 21 day washout period, the subject will then receive Artemether-lumefantrine combination alone for 3 days, with PK sampling at steady state.
  Interventions: Drug: Dolutegravir 50mg od; Drug: Artemether-lumefantrine combination
- Study B Sequence 1 (Experimental): Administration of artesunate-amodiaquine for 3 days with PK sampling at steady state
  Interventions: Drug: Artesunate-amodiaquine
- Study B Sequence 2 (Experimental): Dolutegravir alone for 7 days with PK sampling at steady state, followed immediately by administration of both artesunate-amodiaquine and dolutegravir together for a further 3 days with PK sampling at steady state
  Interventions: Drug: Dolutegravir 50mg od; Drug: Artesunate-amodiaquine

INTERVENTIONS:
Drug: Dolutegravir 50mg od — Dolutegravir 50mg once daily will be given either alone or in combination, as specified
  Other Names: Tivicay, ViiV Healthcare; GSK1349572
  Arms: Study A Sequence 1; Study A Sequence 2; Study B Sequence 2
Drug: Artemether-lumefantrine combination — Artemether-lumefantrine combination will be given both alone and in combination with Dolutegravir 50mg od in order to assess changes in PK
  Other Names: Co-artem
  Arms: Study A Sequence 1; Study A Sequence 2
Drug: Artesunate-amodiaquine — Artesunate-amodiaquine will be given alone or in combination with Dolutegravir 50mg od (in a parallel study design) in order to assess the potential interaction causing changes in PK parameters
  Other Names: Coarsucam
  Arms: Study B Sequence 1; Study B Sequence 2

SUMMARY:
Malaria and HIV are found in the same regions of the world and developing countries are most affected by both diseases. For malaria, new drugs have been introduced called ACTs. These drugs are effective against malaria but little is known about how the levels of these drugs in blood relate to how effective these drugs are. For HIV, a new drug has been developed called dolutegravir which has potential to be widely used in developing countries. This proposal will explore how dolutegravir affects the drug levels of these antimalarial drugs and vice versa. In total, 46 healthy volunteers will participate in this study.

DETAILED DESCRIPTION:
More than 90% of the malaria occurs in sub-Saharan Africa (WHO 2008), the region bearing 67% of the global HIV burden (WHO 2011). Given the extensive overlap in geographical distribution of these diseases, interactions between them could have profound public health consequences. Significant biological interactions exist between HIV and malaria. HIV is known to increase susceptibility to malaria infection (Whitworth, Morgan et al. 2000), compromise the host's ability to clear malaria parasites (characterised by higher parasite densities) (Francesconi, Fabiani et al. 2001), increase the risk of symptomatic malaria and contribute to malaria treatment failure (Hewitt, Steketee et al. 2006). In areas of unstable transmission, malaria mortality is higher in HIV-positive individuals. Additionally, placental malaria infection in HIV positive individuals is associated with higher perinatal mortality, low birth weight and HIV transmission, and this effect is not attenuated in subsequent pregnancies, in contrast with HIV-negative individuals. Conversely, malaria infection has been shown to increase HIV viral load (Hoffman, Jere et al. 1999, Kublin, Patnaik et al. 2005), with the potential for both accelerated HIV disease progression and increased HIV transmission (Abu-Raddad, Patnaik et al. 2006).

As of September 2011, Uganda had 1.4 million people living with HIV/AIDS; of those with clinically advanced disease, 54% (313 117) were receiving ART (WHO). As southern African countries are scaling up coverage of ART, they have also stepped up the fight against Pf malaria by increasing the coverage of Insecticide Treated Nets and by adopting the use of artemisinin-based combination therapies (ACTs) as first line treatment of malaria (USAID 2011). AL and AS-AQ are the most commonly utilized regimens in sub-Saharan Africa for first line treatment for malaria (WHO 2008).

As a consequence of high rates of HIV-malaria co-infection and increasing availability of both ACTs and ART in southern Africa, progressively more co-infected people will receive both classes of drugs. However, the pharmacokinetics, safety and/or efficacy of ACTs such as AL, AS-AQ and DHA-piperaquine in HIV-infected individuals who are on ART are poorly understood. Many efficacy studies conducted as part of the drug development process of ACTs have either not assessed the HIV status of study participants or systematically excluded HIV-infected individuals. Few studies have systematically evaluated for potential drug-drug interactions in a healthy volunteer setting.

Study Design

Open label, fixed sequence healthy volunteer study to compare pharmacokinetic interactions between DTG and AL (Study A; crossover design), or AS-AQ (Study B; parallel group design). Whilst a cross-over study design would be theoretically ideal for investigating both ACTs in combination with DTG, desethylamodiaquine, an active metabolite of AQ has an extensive terminal t1/2 of approximately 10 days; therefore it is not considered feasible to undertake a cross-over design for this arm of the study, since the washout period between the two phases would exceed two months, risking subject attrition. Furthermore, during that time period, intercurrent illnesses and other important changes may occur within a subject, leading changes in eligibility for the study. Therefore, two study designs are planned as detailed in the Study Design Section.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the participant has been informed of all pertinent aspects of the study.
2. Participants who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Men and women aged 18 years and above
4. Weight ≥40 kg
5. HIV antibody negative at screening.
6. Malaria blood film negative at screening
7. Willing to use mosquito bednets routinely for the duration of the study
8. Women of childbearing potential must be willing to use an effective barrier contraception method for the duration of the study.

Exclusion Criteria:

1. Significant disease affecting cardiac, respiratory, gastrointestinal or neurological symptoms which in the clinician's medical judgment could be worsened by participating in this study or the presence of medical or surgical conditions which could prevent the subject from complying with study procedures.
2. Serum alanine transaminase (ALT) levels above 3x upper limit of normal
3. Serum creatinine levels above 2x upper limit of normal
4. Hepatitis B surface antigen positive
5. Use of medications which are known inducers/inhibitors of CYP or glucuronyl transferase UGT1A1 within past 2 months (e.g. anticonvulsants, TB medications, HIV agents for prophylaxis, azole antifungals)
6. Evidence of QT prolongation on electrocardiogram (ECG) QTc (Rate adjusted QT interval) >450ms (men) or >470ms (women)
7. Pregnant women or female subjects who are unwilling to use a suitable contraceptive method for the duration of the study (condom, diaphragm, IUD or contraceptive implant)
8. Likely to be poorly adherent based on clinician's medical judgement
9. Known to be current injection drug user

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2015-06; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change in area under time-concentration curve [AUC] of DTG and antimalarial drugs | At steady state (after 3 days dosing for antimalarials and 7 days for DTG)
  When subjects are at steady state (of single drug or combination, as detailed in the study design section) intensive PK sampling will be performed
Change in maximum concentration [Cmax] of DTG and antimalarials | At steady state (3 days for antimalarials and 7 days for DTG)
  PK sampling will be done when each drug is at presumed 'steady state'
Change in time to maximum concentration [Tmax] for antimalarials and DTG | At steady state (3 days for antimalarials and 7 days for DTG)
  Medications will be dosed up to steady state before PK sampling is undertaken
Change in clearance [Cl/F] for antimalarials and DTG | Steady state - 3 days for antimalarials and 7 days for dolutegravir
  Medications will be dosed up to steady state prior to PK sampling
Change in trough concentration [Ctrough]) for antimalarial drugs and DTG | Steady state - 3 days for antimalarials and 7 days for DTG
  PK sampling will be performed at steady state

SECONDARY OUTCOMES:
Safety and tolerability of the drug combinations | Until 2 weeks after all medication has been discontinued at the end of study
  Patients will be assessed clinically to identify safety concerns, panels of 'safety bloods' will be performed at the time of rich PK sampling, and 12 lead ECGs will assess potential effects of the drugs/ combinations on the QT interval

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed Lamorde, PhD, MBChB, Study Director — Infectious Diseases Institute; Saye H Khoo, FRCP, PhD, Principal Investigator — University of Liverpool
Locations (1):
- Infectious Diseases Institute, Kampala, Uganda

REFERENCES:
- [Derived] Walimbwa SI, Lamorde M, Waitt C, Kaboggoza J, Else L, Byakika-Kibwika P, Amara A, Gini J, Winterberg M, Chiong J, Tarning J, Khoo SH. Drug Interactions between Dolutegravir and Artemether-Lumefantrine or Artesunate-Amodiaquine. Antimicrob Agents Chemother. 2019 Jan 29;63(2):e01310-18. doi: 10.1128/AAC.01310-18. Print 2019 Feb. PMID 30420479
- See also: Dolutegravir product information — https://www.viivhealthcare.com/media/58599/us_tivicay.pdf